CLINICAL TRIAL: NCT01321047
Title: Phase 4 Study of Balanced Propofol Sedation Versus Propofol Alone Sedation
Brief Title: Balanced Propofol Sedation Versus Propofol Alone Sedation in Therapeutic Endoscopic Retrograde Cholangiopancreatography (ERCP)
Acronym: ERCP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Tae Hoon Lee, Soonchunhyang University College of Medicine, Cheonan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCH-2011-18
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Conscious Sedation Failure During Procedure
Keywords: sedation; benzodiazepine; opioid; propofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol group (Active Comparator): the conventional propofol group (P group), sedation was induced by an intravenous bolus injection of propofol (0.5 mg/kg body weight; 10 mg if age > 70 or ASA class III-IV).
  Interventions: Drug: Propofol
- BPS group (Active Comparator): the balanced propofol sedation group (BPS group), both midazolam (0.05 mg/kg body weight; 1 mg if age > 70 or ASA class III-IV) and fentanyl (50 µg; 25 µg if age > 70 or ASA class III-IV) were given intravenously at the initiation of sedation. Thereafter, an initial bolus of propofol (0.5 mg/kg body weight) was given intravenously. Sedation was maintained with repeated doses of 10 to 20 mg propofol.
  Interventions: Drug: BPS

INTERVENTIONS:
Drug: Propofol — propofol (0.5 mg/kg body weight; 10 mg if age > 70 or ASA class III-IV)
  Other Names: A GROUP
  Arms: Propofol group
Drug: BPS — midazolam (0.05 mg/kg body weight; 1 mg if age > 70 or ASA class III-IV) fentanyl (50 µg; 25 µg if age > 70 or ASA class III-IV) propofol (0.5 mg/kg body weight)
  Other Names: B GROUP
  Arms: BPS group

SUMMARY:
Based on previous results, the investigators considered that sedation quality, complications, and procedure outcomes may not be different, however, propofol alone titration may have a fast recovery time than BPS and cost-effectiveness than balanced propofol sedation (BPS). In present study, the investigators therefore evaluate the time and sedation quality of patient recovery, cost-effectiveness, complication, and procedure outcomes between propofol alone and BPS in therapeutic endoscopic retrograde cholangiopancreatography (ERCP).

DETAILED DESCRIPTION:
Previous studies have shown that propofol is superior to traditional sedation regimens with benzodiazepines plus opioids in ERCP procedures. Propofol is a potent hypnotic drug with a short duration of action and consequently a more rapid recovery time for the patients compared with the available Benzodiazepines. Several prospective studies have shown that balanced propofol sedation (BPS) can be used safely and effectively for diagnostic endoscopy under the direction of a gastroenterologist. BPS which was originally described by Cohen et al, combines small incremental doses of propofol with single induction doses of benzodiazepines and opioids under the direction of a physician that is not an anesthesiologist. Because BPS usually targets moderate sedation, adequate amnesia and analgesia can be achieved with concomitant administration of benzodiazepines and opioids. It may cause synergism between propofol and midazolam and reduce dose of propofol. However, there was no proven benefit between propofol alone titrated to moderate level of sedation and BPS; propofol titration combination with benzodiazepines and fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* candidates for therapeutic ERCP

Exclusion Criteria:

* patient age < 18 years
* pregnant women
* inability to provide informed consent
* patients with total gastrectomy
* American Society of Anesthesiologist (ASA) Class V patients
* patients with known respiratory disease, patients with neurologic impairment
* patients with known allergy to the drugs used, history of complications with previous sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Recovery time and cost-effectiveness | SIX MONTH
  Following therapeutic ERCP,full recovery time scoring by Aldrete scoring system and cost measured.

SECONDARY OUTCOMES:
Sedation efficacy, procedure-related outcomes, and complications. | SIX MONTH
  Sedation efficacy parameters was defined as follows; Onset of effective sedation, Patient cooperation (endoscopist, observer-nurse), recovery time, and Patient tolerance (rated by the patients 4hr after procedure).
  Quality of procedure was assessed by procedure outcomes and procedure related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hoon Lee, MD, Study Chair — Soonchunhyang University College of Medicine